CLINICAL TRIAL: NCT01260935
Title: A Prospective Randomized Single-Blinded Multi-Institutional Study Comparing the Laparoscopic Hill and Laparoscopic Nissen Anti-Reflux Procedures
Brief Title: Comparison of Laparoscopic Hill and Laparoscopic Nissen Anti-Reflux Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR 3722
Record Dates: First submitted 2010-11-30; First posted 2010-12-15 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Gastroesophageal Reflux; Esophageal Reflux; Gastroesophageal Reflux Disease; GERD
Keywords: GERD; laparoscopic surgery; gastroesophageal; reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Laparoscopic Hill
  Interventions: Procedure: Laparoscopic Hill Repair
- Arm B (Active Comparator): Laparoscopic Nissen
  Interventions: Procedure: Laparoscopic Nissen Repair

INTERVENTIONS:
Procedure: Laparoscopic Hill Repair — With the Hill repair, stitches are placed right where the esophagus and stomach meet and attached to muscle tissue that is fixed to the spine.
  Arms: Arm A
Procedure: Laparoscopic Nissen Repair — With the Nissen repair, the upper part of the stomach is wrapped around the esophagus, with some anchoring of the wrap at several locations.
  Arms: Arm B

SUMMARY:
The purpose of this study is to compare the effects (good and bad) of the Laparoscopic Hill anti-reflux procedure with the Laparoscopic Nissen anti-reflux surgical procedure to see whether one is better than the other.

DETAILED DESCRIPTION:
The design is a two-armed prospective single-blinded comparison between the two procedures, performed and randomized independently at the Swedish Medical Center Cancer Institute in Seattle, WA, and at Legacy Health Systems in Portland, OR, in adult patients with uncomplicated gastroesophageal reflux failing medical management. A standardized operative technique for each procedures will be utilized at both institutions, and will include intraoperative manometrics and intraoperative photographic documentation of the gastroesophageal valve, as well as placement of clips at the GE junction to accurately identify its location post-operatively. To eliminate "expertise" bias, the investigator from each institution will participate in up to 50 of the first of each of the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* abnormal levels of gastroesophageal reflux documented by pH monitoring who are failing medical management or are requiring maximal medical therapy for control
* > 18 years of age and < 75 years of age

Exclusion Criteria:

* hiatal hernias measuring > 7 cm
* esophageal body amplitude < 30 or in two or more segments
* < 40% propagated peristaltic waves
* GE junction > 5 cm above the esophageal hiatus
* dense fibrotic esophageal strictures which do not markedly improve with pre-operative medical therapy
* body mass index > 40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Determine whether Laparoscopic Hill repair is as effective as Nissen fundoplication for the treatment of gastroesophageal reflux disease (GERD). | 1 year
  Comparison of these two surgical procedures will be based on pre- and post-surgery quality of life questionnaires, manometry (test that measures muscle pressures in the lower esophagus), pH testing, operative time, early complication rates, and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Aye, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (1):
- Swedish Medical Center Cancer Institute, Seattle, Washington, United States